CLINICAL TRIAL: NCT00630383
Title: Immunoregulation by Controlled Parasite Exposure in Multiple Sclerosis.
Acronym: WIRMS-1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: superceded by another similar study
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08025; WIRMS-Pilot
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Multiple Sclerosis
Keywords: Parasite; Necator; immune regulation; regulatory T cells; foxp3; cytokines; multiple sclerosis; hygiene hypothesis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ASP-1 protein, Necator americanus; Histamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients will receive 25 live hookworm larvae.
  Interventions: Biological: Live Hookworm Larvae
- 2 (Placebo Comparator): Patients will receive 0.01 % histamine solution.
  Interventions: Other: Histamine

INTERVENTIONS:
Biological: Live Hookworm Larvae — 25 live hookworm will be applied to the arm and will infect transdermally. They will be eradicated after 48 weeks.
  Other Names: Hookworm; Necator Americanus
  Arms: 1
Other: Histamine — 0.01% histamine solution is pipetted onto a plaster dressing.
  Arms: 2

SUMMARY:
The aim of the study is to determine whether controlled infection with a clinically safe number of larvae of hookworm results in an immune response that is protective in relapsing MS.

DETAILED DESCRIPTION:
Studies have shown that there may be an inverse relationship between infections with worms including hookworms and inflammatory diseases including multiple sclerosis (MS). This has been explained by a protective immune reaction that is triggered by the hookworm in the body that dampens inflammation. In mice with MS, infections with some mouse worms reduced the inflammation and damage to their brain. The primary purpose of this study is to determine whether people with MS who are exposed to a small number of hookworms will develop this protective immune reaction that may reduce MS disease activity. We also plan to determine the effect of the hookworms on relapses during 1 year study.

A study of people with MS naturally infected with intestinal parasites did show significant protection over 5 years, and the levels of biological markers of the infection and some immune substances triggered by it were similar to the ones we obtained with controlled infection in normal volunteers, allergic and asthmatic peoples. We think the study has a genuine potential to benefit people with MS, and there is known interest in the MS patient community. At the therapeutic doses proposed here, this is an innocuous infection. Natural hookworm infection affects 1 billion people worldwide, often without symptoms unless the parasite load is very high. Our controlled exposure studies have shown good tolerability and safety; the risk of infecting others and auto-infection virtually is nil in Western standard hygiene conditions. Many people with MS when asked stated they would prefer an innocuous infection with microscopic larvae to a man-made product that may have more side effects. If the protective mechanisms are determined these studies may also lead to new ways of treating MS, possibly by selecting only the specific chemical components of the worms and the immune response to them that confer protection.

The increase in MS in the Western world, along with other autoimmune inflammatory diseases and asthma may be attributed to decreased exposure to infections such as gut parasites due to improved hygiene ('the hygiene hypothesis'). In animal models, controlled parasite infections including hookworms and related worms protect against MS-like disease. Parasites have evolved host-specific molecular mechanisms to dampen or condition the excessive immune responses against them and thus survive. These parasites induce regulatory mechanisms including Treg and a novel class of B cells that also dampen immune responses called Breg and were recently shown to improve MS in natural infection. They may suppress a class of lymphocytes that cause most damage in MS, Th17 cells. We will produce, with controlled exposure, a similar response to those associated with protective natural exposure in MS. We have the unique combination of expertise in hookworm biology, controlled parasite exposure and immunology of MS and MS trials and our data from our other human studies indicate this is a safe and tolerable intervention of significant potential.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented multiple sclerosis relapsing remitting or secondary progressive with relapses, according to McDonald's criteria, and an MRI scan consistent with MS according to Fazekas criteria
2. Patients with at least 1 relapse in the last 12 months
3. Patients with EDSS score in the range of 0 to 5.5 at the baseline visit
4. Patients of both genders, age >18 years and < 60 years
5. Women of child bearing potential, (who have a negative pregnancy test) must agree to use methods of medically acceptable forms of contraception during the study.
6. Be able and willing to comply with study visits and procedures per protocol.
7. Understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures performed.

Exclusion Criteria:

No populations at risk of severe illness or death will be included in this study

1. Life expectancy < 6 months.
2. Patient is < 5 years free of malignancy, except treated basal cell skin cancer or cervical carcinoma in situ.
3. Patient with grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)
4. Patients with severe and/or uncontrolled medical condition.
5. Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
6. Anaemia (Hb <10 g/dL for females, <11 g/dL for males)
7. Prior or present evidence of parasitic infection; prior treatment with anti-helminthic drugs
8. Patient with serious medical or psychiatric illness that could potentially interfere with the completion of the study treatment according to this protocol
9. History of poor compliance or history of drug/alcohol abuse, or excessive alcohol consumption that would interfere with the ability to comply with the study protocol,
10. Severe asthma, allergy, other autoimmune disease or any condition that the physician judges could be detrimental to subjects participating in this study; including deviations deemed clinically important from normal clinical laboratory

Previous treatment

1. Treatment with interferon or glatiramer acetate or immunosuppressive drugs within 26 weeks prior to baseline
2. Treatment with bone marrow transplantation, total lymphoid irradiation, monoclonal antibodies, umbilical cord stem cells, AIMSPRO at any time prior to baseline
3. Treatment with corticosteroids or ACTH within 4 weeks prior to baseline
4. Treatment with any investigational agent within 12 weeks prior to baseline

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure is an increase in the percentage from total CD4+ T cells of CD4+CD25+foxp3+ cells. | End of study

SECONDARY OUTCOMES:
The expression of foxp3 mRNA from peripheral blood mononuclear cells (PBMC). | End of study
The percentage from total PBMC of NK and NKT cells (CD3-CD56+ and CD3+CD56+ respectively). | End of study
The percentage from total CD3+ T cells of Tr1 cells (CD3+IL10+ T cells). | End of study
The percentage from total PBMC of B regulatory cells (CD20+IL-10+). | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Cris Constantinescu, MD PhD, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospital NHS Trust, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Background] Bach JF. The effect of infections on susceptibility to autoimmune and allergic diseases. N Engl J Med. 2002 Sep 19;347(12):911-20. doi: 10.1056/NEJMra020100. No abstract available. PMID 12239261
- [Background] Edwards LJ, Constantinescu CS. A prospective study of conditions associated with multiple sclerosis in a cohort of 658 consecutive outpatients attending a multiple sclerosis clinic. Mult Scler. 2004 Oct;10(5):575-81. doi: 10.1191/1352458504ms1087oa. PMID 15471376
- [Background] Steinman L. A brief history of T(H)17, the first major revision in the T(H)1/T(H)2 hypothesis of T cell-mediated tissue damage. Nat Med. 2007 Feb;13(2):139-45. doi: 10.1038/nm1551. PMID 17290272
- [Background] Viglietta V, Baecher-Allan C, Weiner HL, Hafler DA. Loss of functional suppression by CD4+CD25+ regulatory T cells in patients with multiple sclerosis. J Exp Med. 2004 Apr 5;199(7):971-9. doi: 10.1084/jem.20031579. PMID 15067033
- [Background] Fleming JO, Cook TD. Multiple sclerosis and the hygiene hypothesis. Neurology. 2006 Dec 12;67(11):2085-6. doi: 10.1212/01.wnl.0000247663.40297.2d. No abstract available. PMID 17159130
- [Background] Correale J, Farez M. Association between parasite infection and immune responses in multiple sclerosis. Ann Neurol. 2007 Feb;61(2):97-108. doi: 10.1002/ana.21067. PMID 17230481
- [Background] Sewell D, Qing Z, Reinke E, Elliot D, Weinstock J, Sandor M, Fabry Z. Immunomodulation of experimental autoimmune encephalomyelitis by helminth ova immunization. Int Immunol. 2003 Jan;15(1):59-69. doi: 10.1093/intimm/dxg012. PMID 12502726
- [Background] Mortimer K, Brown A, Feary J, Jagger C, Lewis S, Antoniak M, Pritchard D, Britton J. Dose-ranging study for trials of therapeutic infection with Necator americanus in humans. Am J Trop Med Hyg. 2006 Nov;75(5):914-20. PMID 17123987
- [Background] Compston A, Coles A. Multiple sclerosis. Lancet. 2002 Apr 6;359(9313):1221-31. doi: 10.1016/S0140-6736(02)08220-X. PMID 11955556
- [Background] Hotez PJ, Pritchard DI. Hookworm infection. Sci Am. 1995 Jun;272(6):68-74. doi: 10.1038/scientificamerican0695-68. PMID 7761817
- [Background] Falcone FH, Pritchard DI. Parasite role reversal: worms on trial. Trends Parasitol. 2005 Apr;21(4):157-60. doi: 10.1016/j.pt.2005.02.002. PMID 15780835
- [Background] Raine T, Zaccone P, Dunne DW, Cooke A. Can helminth antigens be exploited therapeutically to downregulate pathological Th1 responses? Curr Opin Investig Drugs. 2004 Nov;5(11):1184-91. PMID 15573869
- [Background] Quinnell RJ, Bethony J, Pritchard DI. The immunoepidemiology of human hookworm infection. Parasite Immunol. 2004 Nov-Dec;26(11-12):443-54. doi: 10.1111/j.0141-9838.2004.00727.x. PMID 15771680